CLINICAL TRIAL: NCT00329212
Title: Bioequivalence of Bioactive Markers Between Concentrated Herbal Formula and Traditional Herbal Decoctions in Humans
Brief Title: The Pharmacokinetics Study of Concentrated Herbal Formula and Traditional Herbal Decoctions in Humans
Status: Completed | Type: Observational
Sponsor: Committee on Chinese Medicine and Pharmacy (Other Government)
Other Study IDs: CCMP95-RD-010
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2006-11-15 (Estimated); Status verified 2006-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Bioavailability; Therapeutic Equivalency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: San Huang Xie Jin Tang

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics in humans of San Huang Xie Jin Tang (SHXJT) and evaluate the bioequivalence between herbal concentrate and traditional decoction.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers about 6~8 persons should be aged from 20 to 35 years old with a body weight between 50~80 kg, no marriage and have a healthy body condition.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Y C Hou, Professor, Principal Investigator — School of Chinese Medicine, China Medical University
Locations (1):
- Committee on Chinese Medicine and Pharmacy, Department of Health, Taipei, Taiwan, China